CLINICAL TRIAL: NCT06199297
Title: Atezolizumab Plus Bevacizumab Versus Sintilimab Plus Bevacizumab With Transarterial Chemoembolization and Hepatic Arterial Infusion Chemotherapy in Unresectable Hepatocellular Carcinoma: A Multicenter Real-World Study
Brief Title: Atezolizumab Plus Bevacizumab Versus Sintilimab Plus Bevacizumab With TACE and HAIC in Unresectable Hepatocellular Carcinoma
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Binkui Li, Professor, Sun Yat-sen University
Other Study IDs: B2023-690-01
Record Dates: First submitted 2023-12-28; First posted 2024-01-10 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ABTH: Atezolizumab plus bevacizumab combined with TACE-HAIC
  Interventions: Drug: Atezolizumab combined with Bevacizumab; Procedure: Transcatheter arterial chemoembolization and hepatic arterial infusion chemotherapy
- SBTH: Sintilimab plus bevacizumab combined with TACE-HAIC
  Interventions: Drug: Sintilimab combined with Bevacizumab; Procedure: Transcatheter arterial chemoembolization and hepatic arterial infusion chemotherapy

INTERVENTIONS:
Drug: Atezolizumab combined with Bevacizumab — Atezolizumab 1200 mg IV d1, Q3W, combined with bevacizumab 15 mg/kg IV d1, Q3W treatment, treatment continued until disease progression, development of intolerable toxic reactions
  Groups: ABTH
Drug: Sintilimab combined with Bevacizumab — Sintilimab 200 mg IV d1, Q3W, combined with bevacizumab 15 mg/kg IV d1, Q3W treatment, treatment continued until disease progression, development of intolerable toxic reactions
  Groups: SBTH
Procedure: Transcatheter arterial chemoembolization and hepatic arterial infusion chemotherapy — The chemoembolization process employed 30 mg/m2 of epirubicin and 2-10 mL of lipiodol. This was followed by FOLFOX-based HAIC, including 85 mg/m2 of oxaliplatin, 400 mg/m2 of leucovorin, and an initial bolus of 400 mg/m2 of 5-FU for 2 h, which was then followed by a sustained infusion of 1200 mg/m2 5-FU for 23 h.

SUMMARY:
Systemic therapy is the primary option for managing advanced hepatocellular carcinoma (HCC). The combination of atezolizumab and bevacizumab (A+B) has emerged as the first-choice treatment for advanced HCC(IM brave 150). The ORIENT-32 study, also reported an ORR of 24% for sintilimab plus a bevacizumab biosimilar (S+B) versus 8% for sorafenib, with significantly longer OS and PFS. Based on those therapeutic advantages over sorafenib, both the A+B and S+B regimens were approved as first-line treatment options for advanced HCC in China. These two trials had very similar designs but included different target populations. Our previous studies have demonstrated that a novel treatment approach combining transarterial chemoembolization (TACE) with hepatic arterial infusion chemotherapy (HAIC) has high efficacy in patients with potentially resectable HCC or portal vein tumor thrombus. However, it remains unknown whether combining immune checkpoint inhibitors and macromolecular VEGF-targeted therapy with transvascular local interventions could improve patient prognosis in uHCC.

ELIGIBILITY:
Inclusion Criteria:

* (a) a confirmed diagnosis of uHCC;
* (b) at least one target lesion evaluable by both RECIST 1.1 and mRECIST criteria;
* (c) Child-Pugh Grade A or B.

Exclusion Criteria:

* (a) previous exposure to other anti-cancer treatments;
* (b) diagnosis of any other primary malignancy;
* (c) significant esophageal varices or observable red wale marks;
* (d) a history of severe cardiac, pulmonary, or renal comorbidities;
* (e) incomplete follow-up records.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This retrospective real-world study enrolled patients treated in three medical centers in China, including Sun Yat-sen University Cancer Center, Affiliated Cancer Hospital & Institute of Guangzhou Medical University, and Sun Yat-Sen Memorial Hospital. These patients, diagnosed with treatment-naive uHCC, underwent simultaneous combination TACE-HAIC and A+B or S+B.
Sampling Method: Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
objective response rate，ORR | 24 months
  Evaluated according to the criteria for evaluating efficacy in solid tumors (mRECIST and RECIST 1.1)
progression free survival，PFS | 24 months
  Assessed using the mRECIST criteria, defined as patient survival without tumor progression from the start of randomization to the end of year 2

SECONDARY OUTCOMES:
treatment-related adverse events, TRAEs | 24 months
  incidence rates of treatment-related adverse events during the study
overall survival, OS | 24 months
  Defined as the time from the start of randomization to death from any cause

CONTACTS AND LOCATIONS:
Locations (1):
- Wei He, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No